CLINICAL TRIAL: NCT06293625
Title: Personalising and Refining Neo-adjuvant Chemotherapy in Locally Advanced but Resecable Colon Cancer in the Elderly of 70 Years Old or More Phase III Multicentric Open-label Randomized Controlled Trial
Brief Title: Personalising and Refining Neo-adjuvant Chemotherapy in Locally Advanced but Resecable Colon Cancer in the Elderly of 70 Years Old or More
Acronym: FOxTROT2France
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEPAGE PHRCK 2022-2
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Folfox protocol; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeoAdjuvant Chemotherapy arm (Experimental)
  Interventions: Drug: Folfox; Procedure: Surgery
- Current standard of care (Active Comparator)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Folfox — Folfox chemotherapy (folinic acid, fluorouracil and oxaliplatin) for 6 weeks (3 courses) before surgery.
  Arms: NeoAdjuvant Chemotherapy arm
Procedure: Surgery — Experimental arm: Surgery should take place 21 days after the last dose of neoadjuvant chemotherapy Control arm: upfront surgery as soon as possible

SUMMARY:
Colon cancer (CC) is the 5th most common cancer worldwide. Standard care for locally advanced disease is surgical resection followed by 3-6 months of adjuvant chemotherapy (AC) with oxaliplatin and 5-fluorouracil (OxFp).

Almost all of these patients undergo surgery, but many do not receive AC due to frailty (following surgery). This particularly affects patients over 70, who represent the majority of patients diagnosed with CC.

FOxTROT 2, a trial to test the role of NAC in older patients.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed adenocarcinoma of the colon (or upper rectum if too high for radiotherapy), high-grade dysplasia is not acceptable ,
* Patients with synchronous tumors are eligible, if the most advanced tumor meets the criteria above
* Radiological stage T3/T4 and N0/N1/N2 and M0
* Patient eligible for curative surgery (without the need for of chemotherapy)
* No clinical, radiological and colonoscopy evidence of bowel obstruction
* Age ≥ 70 at the time of registration
* pMMR/MSS tumour status
* Fit to receive 6 weeks (3 courses) of NAC with FOLFOX (either full or 80% of FOLFOX dose) and surgery, as assessed by a colon cancer specialist or geriatric oncologist (if available on site).
* Uracilemia <16 ng/ml.
* Adequate full blood count: WBC >3.0 x109/l; platelets >100 x109/l and neutrophils ≥ 1.5 x x109/l Anaemia (Hb < 10.0 g/dl) is not an exclusion, but should be corrected by transfusion prior to surgery and chemotherapy. If Hb remains low despite transfusions, surgery and chemotherapy can be given according to the decision of the surgical and oncology teams.
* Serum electrolytes: Ca2+ > 2.1 mmol/L, Mg2+ > 0.65 mmol/L, K+> 3.4 mmol/LAdequate renal biochemistry: GFR >50 ml/min as assessed by local standards
* Adequate hepatobiliary function:

  * bilirubin < 1.5 x ULN (Patients with Gilbert's syndrome who have raised bilirubin but otherwise normal liver function tests are eligible for the study if bilirubin < 3 x ULN)
  * AST/ALT < 2.5 x ULN
* Patient able to understand and willing to provide written informed consent for the study
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Any patient for whom radiotherapy is advised by the MDT
* Strong evidence of distant metastases or peritoneal nodules (cM1), However, cases with indeterminate abnormalities should be managed and investigated as per standard local MDT procedures and can be considered for trial entry if the MDT opinion is that these are considered most likely to be benign.
* Peritonitis (secondary to perforated tumour)
* T1-T2
* Serious medical comorbidity, as assessed by leading clinician (such as uncontrolled angina)
* Any other malignant disease within the preceding 5 years with the exception of non-melanomatous skin cancer, carcinoma in situ and early stage disease with a recurrence risk <10%
* Known dMMR/ MSI-H tumour status
* Have a peripheral sensitive neuropathy with functional impairment (≥ grade 2 according to NCI-CTCAE v5.0)
* Recent (within four weeks prior to randomisation) or concomitant treatment with brivudine, sorivudine or their chemically related analogues
* Person under guardianship, curatorship, and safeguard of justice or person deprived of liberty
* Impossibility to undergo the medical follow-up of the trial for geographical, social or psychological reasons
* Known hypersensitivity to the active substance of the trial treatments or to any of the excipients
* Patient with poor nutritional status at appreciation by each clinician
* bone marrow hypoplasia
* Potentially severe infection within1 month before NAC
* Patients who have received live attenuated vaccines (yellow fever, varicella, shingles, measles, mumps, rubella, tuberculosis, rotavirus, influenza) within 1 month before NAC
* Any case of clinically significant active heart disease or myocardial infarction within 6 months,
* Any chronic condition not controlled in the last 6 months: Liver failure, renal failure, respiratory failure,
* QT/QTc interval > 450 msec for men and > 470 msec for women
* Known Pernicious anaemia or other anaemias due to vitamin B12 deficiency

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
DFS (disease Free Survival) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No